CLINICAL TRIAL: NCT01902654
Title: Prevalence of Cardiovascular Risk Factors Between Patients With Knee or Hand Osteoarthritis
Brief Title: Osteoarthritis Cardiovascular Risk Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, Joan Calvet Fontova, Dr, Parc Taulí Hospital Universitari
Other Study IDs: Joan02
Record Dates: First submitted 2013-07-09; First posted 2013-07-18 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-11

CONDITIONS: Osteoarthritis; Cardiovascular Risk Factors; Cardiovascular Disease; Metabolic Syndrome
Keywords: Osteoarthritis; cardiovascular disease
MeSH Terms: conditions — Osteoarthritis; Cardiovascular Diseases; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Knee osteoarthritis: Patients over 50 years who presented to an outpatient rheumatology for 1 year and who had knee osteoarthritis.
  Interventions: Other: Cardiovascular risk factors diagnoses collection.; Other: History of cardiovascular disease; Other: Cardiovascular risk factors association
- Hand osteoarthritis: Patients over 50 years who presented to an outpatient rheumatology for 1 year and who had hand osteoarthritis.
  Interventions: Other: Cardiovascular risk factors diagnoses collection.; Other: History of cardiovascular disease; Other: Cardiovascular risk factors association
- Soft tissue disease: All patients over 50 years who presented during the same period of time of other cohorts, to an outpatient rheumatology and who had soft tissue disease with no other rheumatic condition.
  Interventions: Other: Cardiovascular risk factors diagnoses collection.; Other: History of cardiovascular disease; Other: Cardiovascular risk factors association

INTERVENTIONS:
Other: Cardiovascular risk factors diagnoses collection. — We look over patient medical record and we collect the diagnoses associated with cardiovascular risk factor as hypertension, obesity, dislipidemia and diabetes.
Other: History of cardiovascular disease — In all patient we collect the history of cardiovascular disease.
Other: Cardiovascular risk factors association — We have defined two groups according to grouping of none, 1 or 2 cardiovascular risk factors or 3 or more.

SUMMARY:
We analyze retrospectively the relationship between traditional cardiovascular risk factors as hypertension, obesity, dislipidemia and diabetes and hand or knee osteoarthritis and we compare the results with a control groups of patients with soft tissue disease with no other rheumatologic condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for symptomatic hand or knee osteoarthritis
* All patients referred in the same period for soft tissue disease
* > 50 years old

Exclusion Criteria:

* Any other rheumatologic condition
* secondary osteoarthritis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the rheumatology outpatient for symptomatic hand or knee osteoarthritis or soft tissue disease. Patients were referred by their primary care physician, and all patients were visited in primary care assitance.
Sampling Method: Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cardiovascular risk factors in hand or knee osteoarthritis patients | one month
  We analyze the prevalence of cardiovascular risk factors in a cohort of knne osteoarthritis and in a cohort of hand osteoarthritis. Then we evaluate the prevalence of cardiovascular risk factors in a cohort of soft tissue disease patients. Finally we compare osteoarthritis patients with soft tissue disease patients.

SECONDARY OUTCOMES:
Prevalence of cardiovascular disease in hand or knee osteoarthritis. | one month
  We evaluate the prevalence of cardiovascular disease in the three cohorts, hand osteoarthritis, knee osteoarthritis and soft tissue disease; and we compare them.

CONTACTS AND LOCATIONS:
Overall Officials: jordi Gratacos, MD Ph, Study Director — Hospital Parc Tauli
Locations (1):
- Hospital Parc Tauli Sabadell, Sabadell, Barcelona, Spain